CLINICAL TRIAL: NCT03785340
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Masked, Multicenter, Safety and Efficacy Study of Brimonidine Tartrate 0.2% Nanoemulsion Eye Drops in Patients With Dry Eye Disease (DED)
Brief Title: Study of Brimonidine Tartrate Nanoemulsion Eye Drop Solution in the Treatment of Dry Eye Disease (DED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCU-310-301
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye
Keywords: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OCU-310 (Experimental): Brimonidine Tartrate Nanoemulsion Eye Drops 0.20% given 2 times a day for 4 weeks
  Interventions: Drug: Brimonidine Tartrate
- Placebos (Placebo Comparator): Ophthalmic buffered saline Eye Drops given 2 times a day for 4 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Brimonidine Tartrate — Brimonidine Tartrate Nanoemulsion Eye Drops 0.20% given 2 times a day for 4 weeks.
  Other Names: OCU-310
  Arms: OCU-310
Drug: Placebos — Ophthalmic buffered saline Eye Drops given 2 times a day for 4 weeks.
  Other Names: Ophthalmic buffered saline solution
  Arms: Placebos

SUMMARY:
This study evaluates the use of Brimonidine tartrate nanoemulsion eye drop solution in the treatment of Dry Eye Disease (DED). Half of participants will receive Brimonidine and half will receive ophthalmic buffered saline (placebo).

DETAILED DESCRIPTION:
Dry eye disease (DED) is a common ocular disorder involving the aberrant production and instability of tear film, which results in damage to the ocular surface and is correlated with symptoms of ocular discomfort.

This study will be a randomized, placebo-controlled, double-masked, multicenter phase 3 study in the United States conducted at approximately 25 centers. Upon meeting the eligibility criteria, enrolled subjects will be randomly assigned in a 1:1 (test:control) fashion to receive either Brimonidine Nanoemulsion Eye Drops 0.20% investigational product (test) or ophthalmic buffered saline (placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Sign and date informed consent form approved by the IRB
3. History of Dry Eye Disease for ≥6 months
4. Demonstrate the following 2 signs of DED in the same eye at Screening and Baseline (Day 1):

   1. Conjunctival staining at ≥3 (out of a possible score of 6 per eye), and
   2. Schirmer test (with anesthesia) at ≥1 to ≤7mm in 5 minutes
5. Symptomatic evidence of DED by having a global symptom score (Overall SANDE) ≥40 mm at Screening and Baseline (Day 1) visit
6. Intraocular pressure (IOP) ≥ 5 mmHg and ≤22 mmHg in each eye
7. Women who satisfy one of the following:

8a. Are of child-bearing potential (WOCP) who are not pregnant or lactating and who are either abstinent or sexually active on an acceptable method of birth control for at least 4 weeks prior to Visit 1 and throughout the study (i.e., until Day 28), OR 8b. Are post-menopausal or have undergone a sterilization procedure

Exclusion Criteria:

1. Allergic to brimonidine or any similar products, or excipients of brimonidine
2. Use of contact lenses within 14 days prior to Screening visit or planned use during study
3. Currently receiving brimonidine or other treatment for glaucoma or ocular hypertension or history of glaucoma surgery.
4. Receiving or have received any experimental or investigational drug or device within 30 days prior to Screening visit
5. Intraocular pressure <5 mmHg or >22 mmHg in either eye
6. Active ocular infection or history of ocular herpetic keratitis
7. History of neurotrophic keratitis or ocular neuropathic pain
8. Any history of eyelid surgery or intraocular/ocular surgery within the past 3 months
9. Punctal occlusion within 3 months prior to Screening visit or during study
10. Corneal epithelial defect larger than 1 mm2 in either eye
11. Have active drug/alcohol dependence or abuse history
12. Are neonates, pregnant/lactating women, children, or others who may be considered vulnerable populations
13. Received corticosteroid-containing eye drops within 14 days prior to Screening visit or planned use during study
14. Any change in systemic corticosteroids/immunosuppressives, cyclosporine ophthalmic emulsion 0.05% (Restasis®), cyclosporine ophthalmic solution 0.09% (Cequa™), or lifitegrast ophthalmic solution 5% (Xiidra®) within 30 days prior to Screening visit or planned change during study
15. In the opinion of Investigator or Study Coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops
16. Disease, condition, or disorder that in the judgement of Investigator could confound study assessments or limit compliance to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Aesthetic Eye Care Institute/David Wirta, MD and Associates, Newport Beach, California
  - Martel Medical Eye Group, Rancho Cordova, California
  - Rand Eye Institute, Pompano Beach, Florida
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - Heart of America Eye Care, P. A., Mission, Kansas
  - Ophthalmology Associates, St Louis, Missouri
  - Apex Eye- Kenwood, Cincinnati, Ohio
  - Apex Eye-Montgomery, Cincinnati, Ohio
  - Abrams Eye Center, Cleveland, Ohio
  - Scott and Christie Eyecare Associates, Cranberry Township, Pennsylvania
  - Total Eye Care, Memphis, Tennessee
  - Toyos Clinic, Nashville, Tennessee
  - Midtown Eye Physicans & Associates, Houston, Texas
  - Advanced Laser Vision & Surgical Institute, Houston, Texas
  - Revolution Research, Inc; Lake Travis Eye and Laser Center, Lakeway, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

FDAAA 801 VIOLATIONS:
- Correction Confirmed — The responsible party has corrected the violation. — issued 2022-08-01, released 2022-06-29, posted 2022-08-04
- Violation Identified — Failure to Submit. The entry for this clinical trial was not complete at the time of submission, as required by law. This may or may not have any bearing on the accuracy of the information in the entry. — issued 2022-04-15, released 2020-07-15, posted 2022-04-20

RESULTS

PARTICIPANT FLOW:
Groups:
- OCU-310: Brimonidine Tartrate Nanoemulsion Eye Drops 0.20% given 2 times a day (BID) for 4 weeks
- Placebo: Placebo (ophthalmic buffered saline) Eye Drops given 2 times a day (BID) for 4 weeks
Period: Overall Study
Arm/Group | OCU-310 | Placebo
Started | 126 | 126
Received at Least 1 Study Treatment | 126 | 126
Completed | 123 | 126
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set: All randomized participants who previously signed the informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | OCU-310 | Placebo | Total
Number analyzed (Participants) | 126 | 126 | 252
Age, Continuous [Mean (Full Range); unit: years] | 61.7 [27 to 85] | 62.1 [24 to 85] | 62 [24 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 106 | 105 | 211
  Sex: Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 114 | 115 | 229
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 11 | 30
  White | 101 | 111 | 212
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Weeks (Day 28) in Symptom Assessment in Dry Eye (SANDE) Questionnaire Score
Description: The SANDE questionnaire is a short Visual Analog Scale (VAS) assessment that quantifies both severity and frequency of current dry eye symptoms. The SANDE is comprised of two questions, and each question employs a 100-mm horizontal linear VAS. The measurement of symptom frequency ranges from "rarely" to "all of the time", and the symptom severity from "very mild" to "very severe". Data collected from the SANDE questionnaire was calculated by multiplying the frequency score by the severity score and obtaining the square root. The result is the Overall SANDE score which ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
Time Frame: Baseline, 4 weeks (Day 28)
Population: The Intention-to-treat (ITT) set is the primary analysis set for the efficacy endpoints and includes all randomized participants who have at least one post-baseline efficacy measurement. Here, the overall number of participants analyzed is the number of participants with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | OCU-310 | Placebo
Number analyzed (Participants) | 124 | 124
Score on a scale
  Baseline | 73.0 (13.6) | 72.7 (12.4)
  4 weeks (Day 28) | 56.6 (23.2) | 57.2 (19.8)
  Change from Baseline at 4 weeks (Day 28) | -16.4 (20.9) | -15.5 (19.9)
Statistical Analysis 1: Comparison: OCU-310 vs Placebo; Four endpoints (two primary and two secondary) were to be tested in a fixed sequence, proceeding to the next endpoint until a p-value >0.05 was found. The analysis of the four outcomes employed a repeated measures mixed model with mean change from baseline score at the stated time point as the response with baseline score as a covariate and treatment, visit, and their interaction as fixed effects. The least squares mean difference (OCU 310 - placebo) at the stated time point was tested; Test type: Superiority — The endpoints were tested in a fixed sequence, proceeding to the next endpoint until a p-value >0.05 was found: 1. Change from baseline to 4 weeks (Day 28) in SANDE score 2. Change from baseline to 4 weeks (Day 28) in Lissamine Green conjunctival staining scores 3. Change from baseline to 2 weeks (Day 14) in SANDE score 4. Change from baseline to 2 weeks (Day 14) in Lissamine Green conjunctival staining scores; p = 0.739, Mixed Model Repeated Measures Analysis; Least squares mean difference = -0.844, 95% CI 2-sided [-5.823 to 4.134] — Change from baseline to 4 weeks (Day 28) in SANDE score; OCU-310 vs. Placebo

2. Primary Outcome: Change From Baseline to 4 Weeks (Day 28) in Lissamine Green Conjunctival Staining Scores
Description: Conjunctival staining with Lissamine Green dye (1%; LG) staining in each eye was conducted using the slit lamp. A single drop of 1% Lissamine Green dye was applied to the inferior conjunctival fornix of both eyes. The conjunctivae was examined with the slit lamp at ×10 magnification, using a neutral-density filter. The conjunctiva was graded for each eye from 0 to 3 based on the density of punctate staining in the nasal-bulbar and temporal-bulbar zones. Total scores ranged from 0 (no staining) to 6 (most severe staining) with a lower score representing a more desirable outcome.
Time Frame: Baseline, 4 Weeks (Day 28)
Population: The ITT set is the primary analysis set for the efficacy endpoints and includes all randomized participants who have at least one post-baseline efficacy measurement. Here, the overall number of participants analyzed is the number of participants with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OCU-310 | Placebo
Number analyzed (Participants) | 124 | 124
score on a scale
  Baseline | 4.2 (1.1) | 4.1 (1.0)
  4 Weeks (Day 28) | 3.6 (1.6) | 3.2 (1.3)
  Change from Baseline at 4 Weeks (Day 28) | -0.6 (1.4) | -0.9 (1.1)

3. Secondary Outcome: Change From Baseline to 2 Weeks (Day 14) in SANDE Score
Description: as for outcome 1
Time Frame: Baseline, 2 weeks (Day 14)
Population: The ITT set is the primary analysis set for the efficacy endpoints and includes all randomized participants who have at least one post-baseline efficacy measurement. Here, the overall number of participants analyzed are those evaluable for this Outcome Measure and the Number Analyzed per Row is the number of participants with evaluable data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OCU-310 | Placebo
Number analyzed (Participants) | 124 | 124
score on a scale
  Baseline | 73.0 (13.6) | 72.7 (12.4)
  2 weeks (Day 14): number analyzed (Participants) | 122 | 124
  2 weeks (Day 14) | 61.3 (20.5) | 58.6 (17.5)
  Change from Baseline at 2 weeks (Day 14): number analyzed (Participants) | 122 | 124
  Change from Baseline at 2 weeks (Day 14) | -11.6 (18.3) | -14.1 (16.3)

4. Secondary Outcome: Change From Baseline to 2 Weeks (Day 14) in Lissamine Green Conjunctival Staining Scores
Description: as for outcome 2
Time Frame: Baseline, 2 Weeks (Day 14)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OCU-310 | Placebo
Number analyzed (Participants) | 124 | 124
score on a scale
  Baseline | 4.2 (1.1) | 4.1 (1.0)
  2 Weeks (Day 14): number analyzed (Participants) | 122 | 124
  2 Weeks (Day 14) | 3.8 (1.4) | 3.4 (1.3)
  Change from Baseline at 2 Weeks (Day 14): number analyzed (Participants) | 122 | 124
  Change from Baseline at 2 Weeks (Day 14) | -0.4 (1.2) | -0.7 (1.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent completion, throughout the study, and at early termination (Up to 28 Days)
Arm/Group | OCU-310 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/126
Other Adverse Events (participants affected / at risk) | 0/126 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03785340/Prot_SAP_ICF_000.pdf